CLINICAL TRIAL: NCT01114711
Title: Mapping CNS Changes to Frovatriptan Administration in Acute Treatment of Prodrome or Preventative Treatment of Menstrual Migraine (MM)
Brief Title: Frovatriptan and Menstrual Migraine
Acronym: FROVA
Status: Terminated | Type: Observational
Why Stopped: A sister study using Frova at a 10 mg dose had adverse effects.
Sponsor: Mclean Hospital (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, David Borsook, MD, PhD, Director, Pain and Analgesia Imaging Group, Mclean Hospital
Other Study IDs: 2009-P-001452; 400479 (Other Grant/Funding Number: Endo Pharmaceuticals, Inc.)
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Frovatriptan; Menstrual Migraine
Keywords: Menstrual Migraine; Frova; Imaging; fMRI; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Frovatriptan: All subjects will be taking Frovatriptan tablets within 48 hours prior to the scan session (Visit 2).

SUMMARY:
We are looking for women who suffer from menstrual migraine to participate in a 2-visit migraine brain imaging research study. Our goal is to see how the menstrual migraine brain's pain pathways function when the migraineur has been taking Frovatriptan. During the screening visit (Visit 1) participants will sign the informed consent form, complete questionnaires, meet with the study physician, and have QST (quantitative sensory testing: to determine your pain thresholds for a heat stimulus) performed. For Visit 2's MRI scan, subjects will be asked to lie very still while the scan is occurring. In some parts, they will not have to do anything, while in others they will be asked to rate pain and unpleasantness for brush and thermal stimuli. Participants are compensated for both visits.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Regular Menstrual Phase
* Menstrual Migraine
* No significant medical history (Significant medical history of such as seizure disorder, diabetes, alcoholism, cardiac disease including coronary artery disease, psychiatric problems; drug addiction, respiratory problems, liver disease, etc.)
* No significant medication history, except for migraine
* All patients will be currently taking or have previously taken triptan medications for migraine
* Weight, <285 pounds
* Not claustrophobic
* No contraindication to taking triptans

Exclusion Criteria:

* Age <18
* Significant medical problems (aside from pain before, during and after migraine episodes)
* Positive drug of abuse screen (excluding medications currently prescribed for their clinical condition, e.g. opioids, benzodiazepines, etc.)
* Positive alcohol screen
* Women taking oral contraceptives
* Claustrophobia
* History of dermatological hypersensitivity in the facial area
* Positive history of cardiac problems/ abnormalities seen in EKG at initial screening visit
* Pregnancy
* Sensory loss detected on Quantitative Sensory Testing at screening
* Significant alcohol history (ingestion of 5 or more glasses (> 40 oz) of alcohol per week)
* Metal implants of any type (including dental bridges, crowns, retainers, orthodontic devices e.g. braces, etc.)
* Tattoos containing metallic ink on the neck, shoulders, upper arm and head (which could become heated up in the scanner, and potentially cause blistering or burning)
* Cardiac pacemakers
* Aneurysm clips and other vascular stents, filters, clips or other devices
* Prosthetic heart valves
* Other prostheses
* Neuro-stimulator devices
* Implanted infusion pumps
* Cochlear (ear) implants
* Ocular (eye) implants or known metal fragments in eyes
* Exposure to shrapnel or metal filings (sheet metal workers, welders, and others)
* Other metallic surgical hardware in vital areas
* Use of any of the following medications:
* Propanolol/ Inderol
* SSRI's: citalopram/ Celexa, Lepraxo, paroxetine/ Paxil, fluoxetine/ Prozac, Sarafem, Symbyax, sertraline/ Zoloft, Fluvoxamine/ Luvox
* SNRI's: duloxetine/ Cymbalta, venlafaxine/ Effexor
* triptans: sumatriptan/ Imitrex, naratriptan/ Amerge, zolmitriptan/ Zomig, rizatriptan/ Maxalt, eletriptan/ Relpax, almotriptan/ Axert
* ergotamine type medicines: Bellergal, Cafergot, Ergomar, Wiraine, Migranal/ DHE45, Sansert
* ketoconazole (Nizoral, Fungoral)
* itraconazole (Sporanox)
* ritonavir (Norvir)
* erythromycin (Erythrocin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females who suffer from menstrual migraine who are over the age of 18 and have not yet experienced menopause are the study population.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Borsook, MD, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Neuroimaging Center, McLean Hospital, Belmont, Massachusetts, United States